CLINICAL TRIAL: NCT01061489
Title: Computer-based Sensory-cognitive and Physical Fitness Training in Mild Cognitive Impairment (MCI) and Mild Alzheimer's Disease (AD)
Brief Title: Sensory-cognitive and Physical Fitness Training in Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: University of Ulm (Other)
Responsible Party: Principal Investigator, Iris-Tatjana Kolassa, Prof. Dr. Iris-Tatjana Kolassa, University of Ulm
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WIN-Kol-09
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Mild Cognitive Impairment (MCI); Mild Alzheimer's Disease
Keywords: neuroplasticity; Mild Cognitive Impairment (MCI); Alzheimer; sensory-cognitive training; physical fitness
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- sensory-cognitive training (Experimental)
  Interventions: Other: auditory discrimination training
- physical fitness (Experimental)
  Interventions: Other: physical movement training
- waiting list (control group) (No Intervention)

INTERVENTIONS:
Other: auditory discrimination training — 10-week neuroplasticity-based training (5 days/week, 1 hour each, PC-based), training at home
  Arms: sensory-cognitive training
Other: physical movement training — 10-week training, small groups (2 days/week, 1 hour each) plus homework (3 days/week)
  Arms: physical fitness

SUMMARY:
Age-related cognitive decline is unavoidable. However, recent results of neuroplasticity-based research show that neuroplasticity-based training and physical activity might have the potential to decelerate or even reverse effects of aging and age-related cognitive impairments. Little is known whether these results also apply to pathological processes of aging such as mild cognitive impairment (MCI) and dementia.

This multi-center study aims at investigating efficiency and feasibility of a neuroplasticity-based auditory discrimination training and a physical fitness training for patients suffering from mild cognitive impairment or mild Alzheimer's disease (Mini Mental State Examination, MMSE > 19). Evaluation will include neuropsychological testing, electroencephalography (EEG) and magnetic resonance imaging (MRI) measurements as well as blood and liquor analyses.

ELIGIBILITY:
Inclusion Criteria:

* focus: subjective and/or objective memory complaints with MMSE > 19 (MCI or mild Alzheimer's Disease, with stable medication for at least 3 months)
* mild to moderate depression
* corrected-to-normal hearing and vision
* for MRI: non-magnetic metals inside the body
* right handedness preferred

Exclusion Criteria:

* cognitive impairment/ dementia with MMSE < 20, severe psychiatric or neurological disease (current and lifetime)
* physical health that does not allow physical fitness tests and trainings
* benzodiazepin, tricyclic antidepressants
* for MRI: magnetic metal inside the body, cardiac pacemaker etc.
* for liquor: insufficient blood coagulation, insufficient brain pressure

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in global cognition | pre, post, 3-month follow-up
  Average score of the two component scores "memory" and "attention / executive functions", derived from principal component analysis of 11 cognitive items (Munich verbal memory test (MVGT) encoding, MVGT long delayed free recall, free recall of the Alzheimer's Disease Assessment Scale, working memory in the Everyday Cognition Battery, Trail Making Test A and B, digit span forward and backward, digit-symbol-coding and semantic and phonematic fluency).

SECONDARY OUTCOMES:
electrophysiological, MRI, blood and liquor correlates | pre, post, 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Iris-Tatjana Kolassa, Prof. Dr., Study Chair — Clinical and Biological Psychology, University of Ulm
Locations (2):
- Germany (2):
  - University of Konstanz, Konstanz
  - University of Ulm, Memory Clinic, Ulm

REFERENCES:
- [Derived] Kuster OC, Fissler P, Laptinskaya D, Thurm F, Scharpf A, Woll A, Kolassa S, Kramer AF, Elbert T, von Arnim CA, Kolassa IT. Cognitive change is more positively associated with an active lifestyle than with training interventions in older adults at risk of dementia: a controlled interventional clinical trial. BMC Psychiatry. 2016 Sep 8;16(1):315. doi: 10.1186/s12888-016-1018-z. PMID 27608620
- See also: Related Info — http://www.haw.uni-heidelberg.de/forschung/win-neuroplastizitaet.de.html